CLINICAL TRIAL: NCT00050648
Title: Use of Humanized CD25 (Anti-TAC) Monoclonal Antibody and Cyclosporine for the Treatment of Active Psoriasis.
Brief Title: To Study the Effects of CD25 and Low Dose Cyclosporin in the Treatment of Active Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Facet Biotech (Industry)
Responsible Party: James G. Krueger, MD, PhD, Rockefeller University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JKR-0336
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Psoriasis
Keywords: psoriasis; Daclizumab; Cyclosporin; anti-TAC; dermatology; skin
MeSH Terms: conditions — Psoriasis | interventions — Daclizumab; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cyclosporine (Active Comparator): oral medication 2mg/kg/day orally from Day 0 until Day 90
  Interventions: Drug: Cyclosporine
- anti-TAC (Active Comparator): 1mg/kg/dose medication every other week on the odd week (week 1-13)
  Interventions: Drug: Daclizumab
- Cyclosporine and anti-TAC (Experimental): DaclizumabTM at 1mg/kg plus low dose cyclosporine (2 mg/kg/day)
  Interventions: Drug: cyclosporine and Daclizumab

INTERVENTIONS:
Drug: Daclizumab — 1mg/kg medication every other week on the odd week (week 1-13).
  Arms: anti-TAC
Drug: Cyclosporine — 2mg/kg/day orally from Day 0 until Day 90 or a total of 13 weeks.
  Other Names: Neoral
  Arms: cyclosporine
Drug: cyclosporine and Daclizumab — 1mg/kg plus low dose cyclosporine (2 mg/kg/day)
  Arms: Cyclosporine and anti-TAC

SUMMARY:
This study compares the efficacy and analyzes the cellular effects of anti-TAC (Daclizumab) and Cyclosporine in the treatment of psoriasis vulgaris. This is a three-armed study-Daclizumab alone, Cyclosporine alone, and the combination of both Daclizumab and Cyclosporine.

DETAILED DESCRIPTION:
The purpose is to study the safety and effectiveness of a new drug called "anti-TAC" (anti-CD25) Monoclonal Antibody used together with low dose Cyclosporine in the treatment of psoriasis. While the exact cause of psoriasis is unknown, it is believed to involve white blood cells called lymphocytes, which become activated in the skin. It is believed that these activated cells are responsible for the changes you see as the rash of psoriasis. Anti-TAC (anti-CD25) Monoclonal Antibody is designed to block the activation of these lymphocytes. Because the anti-TAC (anti-CD25) Monoclonal Antibody targets the specific cells involved in the symptoms of psoriasis, this new drug may be a better way to treat psoriasis. The second drug, Cyclosporine, is an FDA-approved drug in the treatment of psoriasis. There is evidence in the laboratory that Cyclosporine and anti-TAC, used together, will have an additive effect. An additional benefit of this study is that we are using a lower dose of cyclosporine than is usually given when it is used alone because it is being used together with anti-TAC. This should reduce the side effects usually seen with higher doses of Cyclosporine when it is used as a single drug for psoriasis. The purpose of this study is to test the safety and effectiveness of anti-TAC (Monoclonal Antibody and low dose cyclosporine in patients with active, moderate to severe psoriasis vulgaris. We also hope to gain more information on how anti-TAC works in the body

ELIGIBILITY:
Inclusion criteria

1. Male or female patients with chronic psoriasis vulgaris (disease stable or worsening for > 6 months). Patients age 16 - 21 will be considered on a case by case basis. Patients below 18 will need parental consent.
2. Extensive skin involvement.
3. Scale, thickness, and erythema in individual psoriasis lesions of at least intensity.
4. Psoriasis treated with emollients only for 2 weeks prior to treatment
5. Patients with active psoriatic arthritis, if accompanied by psoriasis vulgaris involving more than 5% of the body surface.
6. History of psoriasis that cannot be treated with topical agents or with previous systemic/ photo(chemo)therapy agents.

Exclusion Criteria:

1. . Positive serology for HIV, Hepatitis B, or Hepatitis C.
2. . Positive β-HCG titer. For women of childbearing potential, unwillingness or inability to use a contraceptive device during this study if negative for β-HCG.
3. Guttate psoriasis, pustular psoriasis, or whole body erythroderma.
4. Active infection or persistent fever of unknown origin. 5.) Major concurrent illness, which could worsen following treatment with DaclizumabTM.

6) Any history of an un-treated neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1997-10; Primary Completion 2004-09 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
clinical tolerability of DaclizumabTM and the DaclizumabTM/cyclosporine combination | day 1, week 1, 2, 3, 4, 5,7,8,9,11, 12, 13, 14

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD, PHD, Principal Investigator — Rockefeller University
Locations (2):
- United States (2):
  - Rockefeller University Hospital, New York, New York
  - Rockefeller University, New York, New York